CLINICAL TRIAL: NCT03765177
Title: Canadian-Led Immunotherapies in Cancer: CLIC-1901 for the Treatment of Patients With Relapsed/Refractory CD19 Positive Hematologic Malignancies
Brief Title: CLIC-1901 for the Treatment of Patients With Relapsed/Refractory CD19 Positive Hematologic Malignancies
Acronym: CLIC-01
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIC-01 Study
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Acute Lymphoblastic Leukemia; Non-Hodgkin's Lymphoma; Chronic Lymphocytic Leukemia
Keywords: Chimeric Antigen Receptor T cells; CLIC-1901; anti-CD19 CAR-T cells
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CLIC-1901 (Experimental): A single Intravenous infusion of CLIC-1901 will be given.
  Interventions: Biological: CLIC-1901

INTERVENTIONS:
Biological: CLIC-1901 — Participants will undergo (a) lymphodepletion with cyclophosphamide and fludarabine, followed by (b) infusion of autologous CLIC-1901 CAR-T cells. All treatments will be delivered intravenously.
  Other Names: autologous anti-CD19 CAR-T cells

SUMMARY:
The investigators propose an early phase study defined as a phase I/II trial assessing safety, feasibility and efficacy of CLIC-1901 autologous anti-CD19 Chimeric Antigen Receptor T cells (CAR-T) cells for participants with relapsed/refractory CD19 positive (CD19+) Acute Lymphoblastic Leukemia (ALL) and non-Hodgkin's Lymphoma (NHL). The Initial Stage of the study (n=20 participants) will focus on feasibility and safety while the Extended Stage will include all participants enrolled in the study (n=additional 80 participants for a total of 100) and will focus on efficacy and safety outcomes. In the proposed trial, we will administer our CAR-T cell product to these participants as a single infusion. Participants will undergo (a) lymphodepletion with cyclophosphamide and fludarabine, followed by (b) infusion of autologous CLIC-1901 CAR-T cells. All treatments will be delivered intravenously.

DETAILED DESCRIPTION:
The investigators have designed a two-stage, single-arm, open-label early phase study to determine the safety and efficacy of CLIC-1901 cell therapy in patients with CD19+ ALL and NHL. The primary objective in the initial stage of 20 participants will be to evaluate the feasibility of our protocol and the safety and tolerability of infusing autologous CLIC-1901 cells into patients with relapsed/refractory CD19+ ALL or NHL. Once 20 participants have been treated and the treatment is deemed safe, up to 80 more participants will be enrolled in an extension stage where the primary objective will be overall response rate (defined as complete or partial response) at 6 months after CLIC-1901 infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have relapsed or refractory CD19+ disease as defined by one of the following:

   a. Relapsed or refractory acute lymphoblastic leukemia or chronic lymphocytic leukemia as defined by one of the following: i. Second or greater relapse ii. Any relapse after allogeneic stem cell transplantation (SCT) iii. Chemorefractory as defined by not achieving CR after 2 cycles of a standard induction chemotherapy or one cycle of salvage therapy b. Histologically confirmed B-cell non-Hodgkin's lymphoma including but not limited to diffuse large B-cell lymphoma (DLBCL) not otherwise specified, primary mediastinal large B-cell lymphoma, or transformed follicular lymphoma, Richter's, Burkitt's or Mantle Cell lymphoma with one of the following: i. Second or greater relapse ii. Any relapse after autologous or allogeneic SCT iii. Chemorefractory as defined by not achieving CR after 2 cycles of a standard chemotherapy or one cycle of salvage therapy
2. All eligible participants must have documentation of CD19 tumour expression demonstrated in tissue biopsy, bone marrow or peripheral blood within the 3 months prior to study screening.
3. Adequate organ function
4. Participant age: 18 to 75 years.
5. Provide written informed consent

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Isolated extra-medullary disease.
2. Participants with concomitant genetic syndrome, such as Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known familial bone marrow failure syndrome.
3. Prior malignancy, except carcinoma in situ of the skin or cervix treated with curative intent and with no evidence of active disease.
4. Prior treatment with any gene therapy product.
5. Participants with polymerase chain reaction (PCR) positive hepatitis B, hepatitis C, or Human Immunodeficiency Virus (tested within 8 weeks of screening), or any uncontrolled infection at screening.
6. Presence of active Graft Versus Host Disease requiring systemic therapy.
7. Participants who have undergone allogeneic SCT less than 6 months prior to CLIC-1901 cell infusion or who have undergone donor lymphocyte infusion less than 6 weeks prior to CLIC-1901 cell infusion.
8. Active Central Nervous System (CNS) involvement by malignancy, defined by CNS-3 per National Comprehensive Cancer Network guidelines.
9. History of anaphylaxis to gentamicin or its derivatives.
10. Participant has received an investigational agent within the 30 days prior to enrolment visit.
11. Pregnant or nursing women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-16 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2042-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants experiencing either Grade 3 or 4 cytokine release syndrome. | Within the first 28 days of CAR-T infusion
  Grade 3 or 4 neurological toxicity, other Grade 3 or 4 toxicity (by CTCAE 4.03) or non-relapse related death.
Proportion of participants with complete (CR) or partial response (PR) to CLIC-1901 | 6 months after CAR-T cell infusion
  Complete response, partial response and disease progression reviewed 6 months after CAR-T cell infusion
Meeting enrollment targets | First 20 participants within 12 months and next 80 participants within 4 years of opening the second stage.
  The feasibility outcome has been met 20 participant in 12 months - currently in next phase and on track to finish on or before October 2024

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Kekre, MD, Principal Investigator — Ottawa Hospital Research Isntitute
Locations (3):
- Canada (3):
  - Vancouver General Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Ottawa Hospital - General Campus, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kekre N, Hay KA, Webb JR, Mallick R, Balasundaram M, Sigrist MK, Clement AM, Nielsen JS, Quizi J, Yung E, Brown SD, Dreolini L, Waller DD, Smazynski J, Gierc NS, Loveless BC, Clark K, Dyer T, Hogg R, McCormick L, Gignac M, Bell S, Chapman DM, Bond D, Yong S, Fung R, Lockyer HM, Hodgson V, Murphy C, Subramanian A, Wiebe E, Yoganathan P, Medynski L, Vaillan DC, Black A, McDiarmid S, Kennah M, Hamelin L, Song K, Narayanan S, Rodrigo JA, Dupont S, Hawrysh T, Presseau J, Thavorn K, Lalu MM, Fergusson DA, Bell JC, Atkins H, Nelson BH, Holt RA. CLIC-01: Manufacture and distribution of non-cryopreserved CAR-T cells for patients with CD19 positive hematologic malignancies. Front Immunol. 2022 Dec 19;13:1074740. doi: 10.3389/fimmu.2022.1074740. eCollection 2022. PMID 36601119
- [Derived] Castillo G, Lalu M, Asad S, Foster M, Kekre N, Fergusson D, Hawrysh T, Atkins H, Thavorn K, Montroy J, Schwartz S, Holt R, Broady R, Presseau J; GO CART team. Hematologists' barriers and enablers to screening and recruiting patients to a chimeric antigen receptor (CAR) T cell therapy trial: a theory-informed interview study. Trials. 2021 Mar 25;22(1):230. doi: 10.1186/s13063-021-05121-y. PMID 33766105
- [Derived] Castillo G, Lalu MM, Asad S, Foster M, Kekre N, Fergusson DA, Hawrysh T, Atkins H, Thavorn K, Montroy J, Schwartz S, Holt RA, Broady R, Presseau J. Navigating choice in the face of uncertainty: using a theory informed qualitative approach to identifying potential patient barriers and enablers to participating in an early phase chimeric antigen receptor T (CAR-T) cell therapy trial. BMJ Open. 2021 Mar 19;11(3):e043929. doi: 10.1136/bmjopen-2020-043929. PMID 33741670
- [Derived] Foster M, Fergusson DA, Hawrysh T, Presseau J, Kekre N, Schwartz S, Castillo G, Asad S, Fox G, Atkins H, Thavorn K, Montroy J, Holt RA, Monfaredi Z, Lalu MM. Partnering with patients to get better outcomes with chimeric antigen receptor T-cell therapy: towards engagement of patients in early phase trials. Res Involv Engagem. 2020 Oct 14;6:61. doi: 10.1186/s40900-020-00230-5. eCollection 2020. PMID 33072399